CLINICAL TRIAL: NCT03095859
Title: Post-operative, Inpatient Rehabilitation After Lung Transplant Evaluation: A Feasibility Study
Brief Title: Post-operative, Inpatient Rehabilitation After Lung Transplant Evaluation
Acronym: PIRATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Benjamin Tarrant, Senior Clinician Physiotherapist - Lung Transplant, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 49/17
Record Dates: First submitted 2017-03-10; First posted 2017-03-30 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Lung Transplant; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Randomized, parallel feasibility trial.
  Stratification as per:
  <55 years of age
  ≥ 55 years
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Single blind study. Treating medical team and therapist delivering standard care will remain blinded to participant allocation. Participants and therapist delivering intensive intervention will be unable to be blinded as they will be receiving / providing intervention. Outcome assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard care (once daily physical rehabilitation, approx. 30 minutes). Standard care will consist of physical exercise, such as early mobility, endurance training, upper limb, lower limb and trunk activity. This will involve non-physical interventions including respiratory therapy, airway clearance and patient and carer education.
  Interventions: Other: Physical rehabilitation.
- Experimental (Experimental): Early intensive physical rehabilitation, which will consist of standard care plus one additional treatment per day. The additional early intensive physical rehabilitation session provided to the experimental group will allow for progression of aerobic, strength and flexibility exercise and / or completion of a more comprehensive physical rehabilitation program.
  Interventions: Other: Physical rehabilitation.

INTERVENTIONS:
Other: Physical rehabilitation. — Early mobility, aerobic exercise, upper and lower limb strength and flexibility training, trunk mobility and core strengthening, inclusive of respiratory therapy and education.

SUMMARY:
This randomized, feasibility trial (n=40) will compare the effects of an intensive, twice daily inpatient physical rehabilitation program against standard care (once daily) following double lung transplantation.

DETAILED DESCRIPTION:
This trial will involve the participation of patients post lung transplantation, in the initial post-operative period. Recruitment will take place as soon as the patient is medically safe and willing to commence physical rehabilitation within the intensive care unit. Current, standard care for inpatient physical rehabilitation post lung transplant involves a once daily session of physiotherapy for the duration of the patient's initial inpatient stay, and consists of early mobility, aerobic exercise, upper and lower limb strengthening and flexibility or core muscle re-training.

This trial aims to assess the feasibility and safety of twice daily physical rehabilitation sessions during the post-operative period following lung transplantation. The content of the additional physical rehabilitation session will not differ from, but will complement current standard care, and will be delivered by a trained research assistant or physiotherapist. To the investigator's knowledge, there is no current evidence to support the dosage and intensity of inpatient physical rehabilitation following lung transplantation, and it is unsatisfactory to use evidence from other patient groups to guide practice in this area.

To assess the feasibility of an intensive, inpatient physical rehabilitation program post lung transplantation, the investigators will collect the following data: Number of patients eligible for study inclusion; number of patients consented; number of additional, intensive physical rehabilitation sessions completed; reasons for non-completion of sessions; and attrition, or patient withdrawal rate. In order to assess the safety of the program, the investigators will also assess for evidence of early, acute rejection of the transplanted lungs based on the routine collection of tissue samples, and adverse events. Adverse events will be defined as any event likely caused by acute physical rehabilitation, including musculoskeletal injury, patient fall and surgical wound breakdown.

These assessments will be complemented by a number of physical and psychological outcome measures and patient statistics, including tests of physical capacity, participation and strength, quality of life, requirements for additional physical rehabilitation and/or hospital readmissions within 10 weeks of study commencement, discharge destination and patient length of stay data. Assessments will be completed within 3 days of first time to mobilize, after three weeks and finally after 10 weeks post-transplant.

The investigators hypothesise that an intensive, physical rehabilitation program will be safe and feasible to implement in the post-operative phase post lung transplantation, and that participants in the intensive rehabilitation group will be more active at 10 days, and at 10 weeks than those receiving standard, post lung transplant physical rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable and able to participate in physical rehabilitation as directed by the treating medical team and primary physiotherapist
* All transplant indications will be included, including re-transplantation
* Will include interstate patients (South Australia, Tasmania) as all patients routinely remain in Victoria attending post-transplant clinic and rehabilitation for three months post operatively

Exclusion Criteria:

* Medically unable to mobilise (e.g. cardiovascular instability)
* Critically unwell (ECMO, CVVHDF etc.)
* <18 years old (paediatric lung transplant)
* Heart-lung transplant
* Single lung transplant (SLTx)
* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Ability to deliver intensive inpatient physical rehabilitation (feasibility). | Patient length of stay is typically two to three weeks following lung transplant surgery.
  Quantified by number of patients eligible for inclusion; number of patients consented; number of additional, intensive physical rehabilitation sessions completed during the initial, inpatient stay post operatively; reasons for non-completion of sessions; and attrition.
  This will be aggregated into an overall percentage of successful delivery of intervention.
Incidence of treatment and non-treatment related adverse events (safety). | Patient length of stay is typically two to three weeks following lung transplant surgery.
  Evidence of early, acute rejection on bronchoscopic biopsy and adverse events. Adverse events will be defined as any adverse outcome during the study period, including but not limited to events that could be related to acute physical rehabilitation such as musculoskeletal injury, patient fall and surgical wound dehiscence or breakdown.

SECONDARY OUTCOMES:
Six-minute walk test. | Pre-transplant results if available. Repeated at 3 and 10 weeks.
  Distance walked in six minutes.
Physical activity monitoring (Dynaport®). | 7 days (5 days of data) at post-operative day 10 and at 10 weeks.
  Physical activity levels.
Pain visual analogue scale (VAS). | Once daily on physical activity monitoring days, from day 10 - 16 post-transplant, repeated for seven days at 10 weeks post-transplant.
  0-10 pain score.
EuroQol EQ-5D-5L. | Baseline (within 3 days from first time to mobilise), 3 weeks and 10 weeks post-transplant.
  Health-related quality of life questionnaire.
Sit to stand test - 60 second. | Baseline (within 3 days from first time to mobilise), inpatient discharge (2-3 weeks), one month and three months.
  Amount of sit-stands completed over 60 seconds.
Grip strength. | Baseline (within 3 days from first time to mobilise), 3 weeks and 10 weeks post-transplant.
  Hand-held dynamometer.
Modified Iowa Level of Assistance Scale (MILOA). | Baseline (within 3 days from first time to mobilise), 3 weeks and 10 weeks post-transplant.
  A valid, reliable and responsive scale of physical capacity in the post-operative patient.

OTHER OUTCOMES:
Length of stay. | Until inpatient discharge, estimated between two to three weeks.
  Length of intensive care and total inpatient stay.
Readmission rates | Inpatient discharge (2-3 weeks) to 10 weeks.
  Readmission rates to the acute setting for the duration of study follow-up.
Discharge destination. | Inpatient (acute) discharge, estimated between two to three weeks.
  Requirement for formal inpatient physical rehabilitation vs home.
Rejection rates. | Baseline to 10 weeks.
  Evidence of any form of chronic lung allograft dysfunction / antibody mediated rejection.
Spirometry | 10 weeks.
  Forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and forced expiratory ratio (FER)).
Adherence to outpatient pulmonary rehabilitation. | Inpatient discharge (2-3 weeks) to 10 weeks.
  Post-transplant outpatient physical rehabilitation uptake - sessions completed.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Tarrant, B.Physio, Principal Investigator — The Alfred
Locations (1):
- The Alfred, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside of this trial.

REFERENCES:
- [Derived] Tarrant BJ, Quinn E, Robinson R, Poulsen M, Fuller L, Snell G, Thompson BR, Button BM, Holland AE. Post-operative, inpatient rehabilitation after lung transplant evaluation (PIRATE): A feasibility randomized controlled trial. Physiother Theory Pract. 2023 Jul 3;39(7):1406-1416. doi: 10.1080/09593985.2022.2041779. Epub 2022 Feb 22. PMID 35193445